CLINICAL TRIAL: NCT04668196
Title: Noninvasive Respiratory Support Outside the Intensive Care Unit in COVID-19 Pneumonia: a Multicentric Study (CATCOVID-AIR)
Brief Title: Noninvasive Respiratory Support in COVID-19 (CATCOVID-AIR)
Acronym: CATCOVID-AIR
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)265/2020
Record Dates: First submitted 2020-12-11; First posted 2020-12-16 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Acute Respiratory Failure; Corona Virus Infection
Keywords: Noninvasive ventilation; High-flow nasal cannula; Severe Acute Respiratory Syndrome; Respiratory Failure; Respiratory Tract Diseases; Coronavirus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Respiratory Insufficiency; Respiratory Tract Diseases | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-flow nasal cannula treatment
  Interventions: Device: High-flow nasal cannula treatment
- Continuous positive airway pressure (CPAP) treatment
  Interventions: Device: Continuous positive airway pressure (CPAP) treatment
- Noninvasive ventilation treatment
  Interventions: Device: Noninvasive ventilation treatment

INTERVENTIONS:
Device: High-flow nasal cannula treatment — Standard operating procedures represented by hihg-flow nasal cannula oxygen therapy
  Groups: High-flow nasal cannula treatment
Device: Continuous positive airway pressure (CPAP) treatment — Standard operating procedures represented by continuous positive airway pressure (CPAP) therapy
  Groups: Continuous positive airway pressure (CPAP) treatment
Device: Noninvasive ventilation treatment — Standard operating procedures represented by noninvasive ventilation treatment
  Groups: Noninvasive ventilation treatment

SUMMARY:
COVID-19 pneumonia can cause severe acute hypoxemic respiratory failure. The usefulness of noninvasive respiratory support (NIRS), by means of nasal high-flow oxygen (NHFO), continuous positive airway pressure (CPAP), or noninvasive ventilation (NIV), established outside the intensive care unit, is unknown. The aim of this multicenter, retrospective, longitudinal study is to compare the effectiveness of these treatments to prevent death or endotracheal intubation at day 28, and what factors, related to the disease or to the characteristics of the treatment itself, can condition its success or failure.

DETAILED DESCRIPTION:
Multicenter, retrospective, longitudinal study in consecutive adult COVID-19 patients with acute respiratory failure, requiring noninvasive respiratory support (NIRS) outside the intensive care unit (ICU) in 10 hospitals in Catalonia (Spain). Demographic, laboratory, clinical and noninvasive respiratory support data will be collected and analyzed according to the primary outcome (death or endotracheal intubation at day 28) and secondary outcomes (see the dedicated section).

During the hospitalization, patients were treated according to the standard procedures of the participating centers. This study is observational and no randomization have been performed.

Patients were followed up to either 28-days or hospital discharge if still hospitalized at day 28 from NIRS initiation.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 pneumonia confirmed with polymerase chain reaction (PCR).
* Acute respiratory failure.
* Treated by noninvasive respiratory support (nasal high-flow oxygen, CPAP or noninvasive ventilation), initiated outside the intensive care unit.
* Age > 18 years

Exclusion Criteria:

* Acute respiratory failure not related to COVID-19
* Hypercapnic acute respiratory failure
* Early intolerance to treatment
* Nosocomial infection
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID19 patients treated by noninvasive respiratory support (nasal high-flow oxygen, CPAP, or noninvasive ventilation), initiated outside the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 28 days within noninvasive respiratory support initiation
  Death or endotracheal intubation

SECONDARY OUTCOMES:
28-day mortality | 28 days within noninvasive respiratory support initiation
Hospital mortality | Until 28 days from noninvasive respiratory support initiation
  Any death during hospital stay
Endotracheal intubation | 28 days within noninvasive respiratory support initiation
Duration of hospital stay | Until 28 days from noninvasive respiratory support initiation
  Time between admission and discharge from hospital or death in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Júlia Sampol, MD, Study Chair — Hospital Universitari Vall d'Hebron Research Institute; Sergi Marti, MD PhD, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Fundació Althaia, Manresa, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Universitari Mútua Terrassa, Terrassa, Bardelona
  - Hospital del Mar, Parc de Salut Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Dr.Josep Trueta, Girona

REFERENCES:
- [Derived] Marti S, Carsin AE, Sampol J, Pallero M, Aldas I, Marin T, Lujan M, Lalmolda C, Sabater G, Bonnin-Vilaplana M, Penacoba P, Martinez-Llorens J, Tarrega J, Bernadich O, Cordoba-Izquierdo A, Lozano L, Mendez S, Velez-Segovia E, Prina E, Eizaguirre S, Balana-Corbero A, Ferrer J, Garcia-Aymerich J. Higher mortality and intubation rate in COVID-19 patients treated with noninvasive ventilation compared with high-flow oxygen or CPAP. Sci Rep. 2022 Apr 20;12(1):6527. doi: 10.1038/s41598-022-10475-7. PMID 35444251